CLINICAL TRIAL: NCT03680859
Title: The NIDDK Gastroparesis Registry 3: Characterization and Clinical Course of Symptoms and Gastric Emptying in Patients With Symptoms of Gastroparesis
Brief Title: Gastroparesis Registry 3
Acronym: GpR3
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Johns Hopkins University (Other); Massachusetts General Hospital (Other); Temple University (Other); University of Louisville (Other); Wake Forest University (Other); Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Sponsor
Other Study IDs: 7 DK GpR3; U01DK073983 (NIH); U01DK112193 (NIH); U01DK073975 (NIH); U01DK074035 (NIH); U01DK074007 (NIH); U01DK073974 (NIH); U24DK074008 (NIH)
Record Dates: First submitted 2018-09-07; First posted 2018-09-21 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Gastroparesis; Diabetic Gastroparesis; Idiopathic Gastroparesis
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, and PBMC specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Diabetic: Participants with a primary etiology of diabetic gastroparesis
- Idiopathic: Participants with a primary etiology of idiopathic gastroparesis
- Post-fundoplication: Participants with a primary etiology of post-Nissen fundoplication gastroparesis
- Diabetic with Normal Emptying: Diabetic participants with symptomatic nausea and vomiting with normal gastric emptying
- Idiopathic with Normal Emptying: Idiopathic participants with symptomatic nausea and vomiting with normal gastric emptying
- Post-fundoplication with Normal Emptying: Post-fundoplication participants with symptomatic nausea and vomiting with normal gastric emptying

SUMMARY:
The purpose of this study is to create a new registry of patients with gastroparesis in order to better understand the characteristics of patients with gastroparesis and follow how their condition changes over time. The data collected may improve the understanding of the condition to enable better diagnosis and treatment.

DETAILED DESCRIPTION:
GpR 3 is an observational study of patients with symptoms of gastroparesis with either delayed or normal gastric emptying. Epidemiological, clinical, physiological, and patient outcome data will be collected to characterize the patients and their clinical course to better understand this disorder. The long-term goal is to help phenotype patients into pathophysiologically defined subsets. This classification will provide a foundation for translational research, facilitating the search for etiopathogenesis and enhance the ability to define and conduct large clinical trials, ultimately leading to the development of more rational and effective therapeutic approaches for gastroparesis.

The primary objectives of the Gastroparesis Registry 3 (GpR 3) are:

* To create a new registry of patients with symptoms of gastroparesis, both patients with delayed gastric emptying and patients with similar symptoms but normal gastric emptying, for the enhanced study of symptoms, gastric motility abnormalities, patient characteristics, and degree of morbidity.
* To follow a well-characterized cohort to further define the natural history and clinical course of patients with symptoms of gastroparesis - both symptoms and gastric emptying over time. Treatments given for their clinical care and clinical responses to treatments will be recorded.
* To provide a reliable source for recruitment of well-characterized patients with gastroparesis for other studies including therapeutic clinical trials, pathophysiological, molecular, histopathologic, or other ancillary studies. These subsequent clinical trials or ancillary studies will be conducted under separate study protocols with separate consent processes.

Specific secondary objectives of GpR3 have been developed to allow the patients entered in GpR3 to help advance our understanding of gastroparesis:

* Assess several areas of gastric motility in patients with symptoms of gastroparesis (fundic accommodation, antral contractility, global gastric emptying).
* Determine the change in gastric motility over time, in patients with gastroparesis and in patients with symptoms of gastroparesis but normal gastric emptying.
* Evaluate the clinical symptomatic course (outcome) of patients followed in the registry.
* Use the registry to better capture clinical treatment responses to specific treatments while patients are in the registry.
* Characterize abdominal pain in patients with gastroparesis and gastroparesis-like syndrome by:

  * Describing the abdominal pain seen in patients with gastroparesis
  * Determining if the pain has neuropathic or nociceptive qualities
  * Determining attributes of patients with abdominal pain
  * Assessing patients in the presence of sensory gastric dysfunction
  * Objective mapping of the abdominal pain and determining central and/or peripheral attributes of the abdominal pain
* Compare the Rome IV categories of gastric disorders (functional dyspepsia (FD), epigastric pain syndrome (EPS), postprandial distress syndrome (PDS), chronic idiopathic nausea and vomiting (CINV), rumination syndrome, cyclic vomiting syndrome, central abdominal pain syndrome) to our present classification of gastroparesis and gastroparesis-like disorder.
* Determine the prevalence of hypermobility spectrum disorders (HSD) in patients with gastroparesis.
* Compare the water load satiety test (WLST) to intragastric meal distribution (IMD) during scintigraphy and to symptoms of early satiety, postprandial fullness in patients with symptoms of gastroparesis.
* Collect serum, plasma, and peripheral blood mononuclear cells (PBMC) that can be used for subsequent analysis to address specific research questions.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of gastroparesis of at least 12 weeks' duration with varying degrees of nausea, vomiting, early satiety, postprandial fullness
* An etiology of either diabetic, idiopathic, or post-fundoplication (Nissen, Dor, or Toupet) gastroparesis or gastroparesis-like disorder (symptoms of gastroparesis but normal gastric emptying)
* Gastric emptying scintigraphy of solids using the 4-hour Egg Beaters® protocol (or equivalent generic liquid egg white meal) within the last 6 months with either:
* Abnormal gastric emptying rate defined as an abnormal 2 hour (>60% retention) and/or 4 hour (>10% retention) result based on a 4 hour scintigraphic gastric emptying study. (This group will comprise ~75% of patients in the registry.)
* Patients with a normal gastric emptying rate, but who have symptoms of gastroparesis. (This group will comprise ~25% of patients in the registry.)
* Negative upper endoscopy or upper radiographic GI series within 2 years of registration
* Age at least 18 years at initial screening visit

Exclusion Criteria:

* Inability to comply with or complete the gastric emptying test by scintigraphy (including allergy to eggs)
* Use of narcotic analgesics greater than three days per week
* Presence of other conditions that could explain the patient's symptoms:
* Pyloric or intestinal obstruction: by EGD, UGI, or Abdominal CT
* Active inflammatory bowel disease
* Known eosinophilic gastroenteritis or eosinophilic esophagitis
* Primary neurological conditions that can cause nausea and vomiting such as increased intracranial pressure, space occupying or inflammatory/infectious lesions
* Acute renal failure
* Chronic renal failure (serum creatinine >3 mg/dL) and/or on hemodialysis or peritoneal dialysis
* Acute liver failure
* Advanced liver disease (Child's B or C; a Child-Pugh-Turcotte (CPT) score of ≥7)
* Prior gastric surgery including total or subtotal (near complete) gastric resection, esophagectomy, gastrojejunostomy, gastric bypass, gastric sleeve, pyloroplasty, pyloromyotomy. Note: patients with prior Nissen, Dor, or Toupet fundoplication will be eligible for enrollment.
* Any other condition, which in the opinion of the investigator, could explain the symptoms or interfere with study requirements
* Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females at least 18 years old at the initial screening interview in the United States who are:
  * Diabetic, idiopathic, or post-fundoplication gastroparesis patients with delayed gastric emptying
  * Diabetic, idiopathic, or post-fundoplication patients with symptoms of gastroparesis but with normal gastric emptying
Sampling Method: Non-Probability Sample
Enrollment: 406 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline GSCI score at 48 weeks | Baseline to 48 weeks
  The outcome is assessed using the self-reported postprandial fullness/early satiety subscore, which is computed as the average of 4 scores for 4-items on the Gastroparesis Cardinal Symptom Index (GCSI) survey: stomach fullness, inability to finish a normal-sized meal, feeling excessively full after meals, and loss of appetite. Each item is scored from 0 (no) to 5 (very severe) symptoms in the past 2-weeks; the subscore ranges from 0 to 5. The change is computed as the subscore at 48-weeks minus the baseline subscore.

SECONDARY OUTCOMES:
Change from baseline in Short Form Health Survey (SF-36v2) physical health QOL component score at 48 weeks | Baseline to 48 weeks
  The outcome is assessed using the self-reported 36-item Short Form Health Survey (SF-36v2) physical health QOL component score. The score ranges from 0 (poorest) to 100 (highest) QOL. The change is computed as the score at 48-weeks minus the baseline score.
Change from baseline in Short Form Health Survey (SF-36v2) mental health QOL component score at 48 weeks | Baseline to 48 weeks
  The outcome is assessed using the self-reported 36-item Short Form Health Survey (SF-36v2) mental health QOL component score. The score ranges from 0 (poorest) to 100 (highest) QOL. The change is computed as the score at 48-weeks minus the baseline score.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Parkman, MD, Study Chair — Temple University Hospital; Braden Kuo, MD, Study Chair — Massachusetts General Hospital; Pankaj J Pasricha, MD, Study Chair — Johns Hopkins University
Locations (6):
- United States (6):
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital-Digestive Healthcare Center, Boston, Massachusetts
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center (TTUHSC), El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Public use complete database will be submitted to the NIDDK Data Repository
Supporting Information: Study Protocol, ICF
Time Frame: Two years after the end of the funding period
Access Criteria: An investigator interested in acquiring GpR3 study data should contact the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Central Repository at https://www.niddkrepository.org/search/study/ and apply to obtain the data required for their study. IRB approval
URL: https://repository.niddk.nih.gov/home/

REFERENCES:
- See also: Gastroparesis Clinical Research Consortium — https://jhuccs1.us/gpcrc/